CLINICAL TRIAL: NCT03473899
Title: A Prospective, Randomized, Double-blind, Placebo Controlled Single Centre Trial to Assess the Efficacy and Safety of rESWT Combined With a Specific Rehabilitation Program for Acute Hamstring Muscle Complex Injury Type 3b in Athletes
Brief Title: Radial Extracorporeal Shock Wave Therapy for Acute Hamstring Muscle Complex Injury Type 3b in Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kinef Kinesiología Deportiva (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CrupnikDolorClastMuscleInjury
Record Dates: First submitted 2018-03-10; First posted 2018-03-22 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Athletic Injuries
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: A medical assistant at the clinic of the Principal Investigator will allocate interventions by means of opaque sealed envelopes that will be marked according to the allocation schedule. The medical assistant will be unaware of the size of the blocks.
  The randomized intervention assignment as outlined above will be concealed from both patients and health care staff until recruitment will be complete and irrevocable.
  Patients will be blinded in this study. The assessor will be blinded in this study. The assessor is the person who will assess the outcome of treatment during follow up. In this study, the assessor will be a medical assistant at the clinic of the Principal Investigator.
  The therapist will not be blinded in this study. The therapist is the person who will administer either rESWT or sham-rESWT to the patient. In this study, the therapist will be the Principal Investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rESWT + RP (Active Comparator): Device: rESWT
  Interventions: Device: rESWT
- sham-rESWT + RP (Placebo Comparator): Device: sham-rESWT
  Interventions: Device: Sham-rESWT

INTERVENTIONS:
Device: rESWT — rESWT will be performed as follows:
  * Nine rESWT sessions
  * Three sessions per week
  * rESWT device: Swiss DolorClast (Electro Medical Systems, Nyon Switzerland), EvoBlue handpiece, 15 mm applicator
  * 2500 rESWs per session, with energy density between 0.12 and 0.16 mJ/mm^2, depending on what the patient tolerates
  * rESWs applied at 15 Hz
  * Application of rESWs in prone position, with the patient lying on an examination table
  * Exact location of the application of rESWs determined by clinical and ultrasonographic examinations
  * Treatment of both the side of injury and the entire affected muscle (from distal to proximal in order to relax the affected muscle)
  * No use of local anesthesia.
  In addition, patients will receive a specific rehabilitation program.
  Arms: rESWT + RP
Device: Sham-rESWT — Sham-rESWT will be performed as rESWT described in Arm rESWT + RP, but with a specially designed placebo EvoBlue handpiece that looks and sounds like the EvoBlue handpiece of the Swiss DolorClast, but does not generate radial shock waves. This is achieved by blocking the projectile shortly before it strikes the metal applicator. The placebo EvoBlue handpiece will not emit any radial shock wave energy.
  In addition, patients will receive a specific rehabilitation program.
  Arms: sham-rESWT + RP

SUMMARY:
This study tests the hypothesis that the combination of radial extracorporeal shock wave therapy performed with the Swiss DolorClast device (Electro Medical Systems, Nyon, Switzerland) and a specific rehabilitation program (hereafter, "rESWT + RP") is effective and safe in treatment of acute hamstring muscle complex injury Type 3b, and is statistically significantly more effective than the combination of sham-rESWT and RP (hereafter, "sham-rESWT + RP").

DETAILED DESCRIPTION:
Acute injuries of the hamstring muscle complex (HMC) are frequently observed in various sports disciplines both in elite and recreational sport, and are the most common injury in soccer. Despite intensive research into prevention and management of acute HMC injury during the last decade epidemiological data show no decline in injury and re-injury rates. In this regard a recent study prospectively observed 374 Danish elite soccer players during a 12-month period and registered 46 first-time and eight recurrent HMC injuries (incidence rates: 12.3% [first-time injuries] and 2% [recurrent injuries]). Statistically significantly more players experienced a first-time acute HMC injury during a match than during training. Moreover, among 32 players who suffered from acute HMC injury in a period of 12 months before the study, eight players incurred an injury that fulfilled the criteria for a recurrent injury (incidence: 25%). Approximately two thirds of the first-time injuries were categorized as moderate, with time to return to play between 8 to 28 days.

Anatomical and functional aspects of the HMC predispose it to injury, including the fact that the muscles cross two joints and undergo eccentric contraction during the gait and running cycle.

Acute HMC injury typically occurs through an eccentric mechanism at the terminal stages of the swing phase of running. The long head of the biceps femoris (LHBF) muscle is most commonly affected, and within the LHBF muscle, the proximal myotendinous junction and proximal locations are most commonly affected.

The diagnosis of acute HMC injury is based on the presence of acute-onset pain in the posterior thigh, and presence of the triad of pain on contraction, stretching and palpation. Imaging has a role in confirming the site of injury and characterizing its extent, providing some prognostic information and helping plan treatment. In this regard both magnetic resonance imaging (MRI) and ultrasonography (US) have been shown to be effective for identification of hamstring strains and tendinopathy. Both MRI and US provide detailed information about the HMC with respect to localization and characterization of injury. Several clinical, MRI and US determinants were established that are associated with a longer recovery time in nonoperative management of acute HMC injury. However, it is important to realize that for an individual HMC injury none of these MRI and US determinants show a direct correlation with the time to return to play. Accordingly, the prognosis of HMC injuries should not be guided by imaging findings alone.

Precise classification of acute HMC injury has important implications for treatment and prognosis (i.e., time to return to play), as outlined in detail below. There are anatomical differences between a Type 3a injury (minor partial muscle tear ≤ 5 mm; intrafascicle/bundle-tear) and a Type 3b injury (moderate partial muscle tear > 5 mm; interfascicle/bundle-tear).

Acute HMC injuries Type 4 (i.e., subtotal or complete muscle tear or tendinous avulsion) require early surgical repair. However, acute HMC injuries Type IV are rare.

The treatment of choice of acute HMC injuries Type 3a and 3b is a progressive physiotherapeutic exercise programme. Besides this, there is currently only insufficient scientific evidence to support other treatment methods, including local infiltrations. In particular, injections of platelet-rich-plasma (PRP) showed no effect when compared to control.

It is of note that another study that was published very recently in the The New England Journal of Medicine demonstrated the negative clinical consequences of protracted immobilization after an acute muscle injury Type 3b in recreational sports. Starting rehabilitation two days after injury rather than waiting for nine days shortened the interval from injury to pain-free recovery and the time to return to play by approximately three weeks without any significant increase in the risk of reinjury. The authors of this study concluded that the observed difference supports the importance of early loading of injured musculotendinous tissue.

Acute muscle injuries Type 3a and 3b have different time frames for recovery and return to play, with optimal treatment between 10 and 14 days in case of Type 3a and on average approximately six weeks in case of Type 3b. However, particularly in case of acute HMC injury Type 3b there is considerable interindividual variability in the time frame for return to play.

Most importantly, particularly the high reinjury rate of acute HMC injury suggests that commonly utilized rehabilitation programs may be inadequate at resolving possible muscular weakness, reduced tissue extensibility, and/or altered movement patterns associated with the injury. Accordingly, there is need for developing innovative treatment options particularly for acute HMC injury Type 3b.

Very recently it was demonstrated that extracorporeal shock wave therapy (ESWT) may accelerate regeneration after acute skeletal muscle injury. The use of extracorporeal shock waves in medicine was first reported over 30 years ago as a treatment for kidney stones, and is commonly referred to as 'extracorporeal shock wave lithotripsy', or 'ESWL'. Extracorporeal shock waves are also used as a treatment for musculoskeletal conditions such as plantar heel pain and boney non-union, and is commonly referred to as 'extracorporeal shock wave therapy' (ESWT) to differentiate from ESWL.

There are three different types of extracorporeal shock waves that could be used in ESWT for acute HMC injury Type 3b, focused, defocused and radial, and several modes of operation of focused, defocused and radial extracorporeal shock wave generators.

To our knowledge randomized controlled trials (RCTs) testing efficacy and safety of rESWT for acute HMC injury Type 3b have not yet been published. In contrast, rESWT has become an established treatment modality for various musculoskeletal conditions such as calcifying tendonitis of the shoulder, tennis elbow and plantar fasciopathy, to mention only a few. Among the 44 RCTs on rESWT currently listed in the PEDro database (status of September 09, 2017), 29 (66%) were performed with the rESWT device Swiss DolorClast (Electro Medical Systems, Nyon, Switzerland).

The investigators of the present study have extensive practical experience with rESWT for various musculoskeletal conditions using the Swiss DolorClast. Most importantly, all of us have already gained practical experience with rESWT for acute HMC injury Type 3b in athletes. One of our most prominent patients was a professional soccer player at a European top club (regularly playing in the UEFA Champions League) who incurred a HMC injury Type 3b and returned to play (full 90-min match with his national team) 35 days later. In the aforementioned studies published in the New England Journal of Medicine the cumulative probability of resumptions of sports activity on day 35 after acute HMC injury Type 3b in professional soccer players or recreational athletes was only respectively 20% or 5% after treatment with a rehabilitation program.

Considering the limited evidence of efficacy and safety of rESWT for acute HMC injury Type 3b, further research is needed to support the use of rESWT for this condition. Taking into account the proven efficacy and safety of rESWT using the Swiss DolorClast for treating musculoskeletal conditions, the widespread use of the Swiss DolorClast based on its proven efficacy and safety, and our own very promising pilot data of rESWT using the Swiss DolorClast for treating acute HMC injury Type 3b in athletes it is reasonable to hypothesize that (i) the combination of rESWT and a specific rehabilitation program is effective and safe in treatment of acute HMC injury Type 3b, (ii) this combination therapy is statistically significantly more effective than the same specific rehabilitation program alone, and (iii) this combination therapy will gain widespread acceptance as soon as effectiveness and safety will be demonstrated in a randomized controlled trial. This is the main purpose of the proposed study.

ELIGIBILITY:
Inclusion Criteria:

* Adults (both male and female) with clinical and ultrasonographic diagnosis of acute HMC injury Type 3b
* Age range: between 18 and 35 years
* Physical conditions for rehabilitation (i.e., no surgery required)
* Willingness of the patient to participate in the study, and written informed consent signed and personally dated by the patient
* No contraindications for rESWT

Exclusion Criteria:

* Children and teenagers below the age of 18
* Adults aged >35 years old
* Patients with clinical and ultrasonographic diagnosis of acute HMC injury Type 3b who got injured more than seven days before potential enrollment into this study
* Patients with clinical and ultrasonographic diagnosis of acute HMC injury Type 3A or Type 4
* Bilateral acute HMC injury (Types 3A, 3B or 4)
* Proven or suspected HMC injury (Types 3A, 3B or 4) of the same lower limb in the time period of six months before potential enrollment into this study
* Muscle injury caused by external impact on the back of the affected thigh
* Surgery on the affected lower limb in the time period of one year before potential enrollment into this study
* Acute or chronic lumbar pathology (because some cases of thigh pain may relate to spinal pathology)
* No willingness of the patient to participate in this study, and/or written informed consent not signed and not personally dated by the patient
* Contraindications of rESWT, i.e., treatment of pregnant patients, treatment of patients with blood-clotting disorders (including local thrombosis), treatment of patients treated with oral anticoagulants, treatment of patients with local bacterial and/or viral infections/inflammations, treatment of patients with local tumors, and treatment of patients treated with local corticosteroid applications in the time period of six weeks before the first rESWT session (if applicable).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-22 (Actual); Primary Completion 2020-03-21 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Individual time (days) necessary to return to play. | From date of randomization until the date of return to play, up to six months
  Individual treatment success is defined as the possibility to return to play, fulfilling all criteria specified by Van de Horst et al. (Sports Med 2016;46(6):899-912). Accodingly, the primary outcome measure is the number of days until "yes" (return to play possible according to the criteria established by Van de Horst et al., 2016) will be achieved.

SECONDARY OUTCOMES:
Individual patient's satisfaction | Six months after randomization
  Individual patient's satisfaction will be assessed using a scale ranging from 0 (maximum dissatisfaction) to 10 (maximum satisfaction)
Presence or absence of re-injury | From date of randomization up to six months
  Re-injury is defined as sudden, sharp pain in the posterior aspect of the thigh that was initially injured, accompanied by the same objective criteria initially used for the diagnosis of acute HMC injury Type 3b

CONTACTS AND LOCATIONS:
Overall Officials: Javier Crupnik, PT, Principal Investigator — Kinef Kinesiología Deportiva
Locations (1):
- KinEf Kinesiología Deportiva, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers.

REFERENCES:
- [Derived] Crupnik J, Silveti S, Wajnstein N, Rolon A, Vollhardt A, Stiller P, Schmitz C. Is radial extracorporeal shock wave therapy combined with a specific rehabilitation program (rESWT + RP) more effective than sham-rESWT + RP for acute hamstring muscle complex injury type 3b in athletes? Study protocol for a prospective, randomized, double-blind, sham-controlled single centre trial. J Orthop Surg Res. 2019 Jul 23;14(1):234. doi: 10.1186/s13018-019-1283-x. PMID 31337441

DOCUMENTS (1):
  • Study Protocol (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT03473899/Prot_000.pdf